CLINICAL TRIAL: NCT06420102
Title: Detecting Changes in Skin Status Over the Site of a Stage 1 Pressure Ulcer Using Biophysical Sensors and Biomarkers
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Collaborators: European Union (Other); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ERGO 66933
Record Dates: First submitted 2023-08-23; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Grade 1 pressure ulcer cohort: Individuals who are in hospital that present with a confirm grade 1 pressure ulcer. These include a range of sex, age and ethnicities.
  Interventions: Diagnostic Test: Biophysical and biochemical skin assessment

INTERVENTIONS:
Diagnostic Test: Biophysical and biochemical skin assessment — Measurements are taken from the skin surface including transepidermal water loss, skin hydration and pH. In addition, non-invasive biofluid (sebum) is sampled from the skin to profile local inflammation. Skin surface cells were also stripped to assess corneocyte properties over the pressure ulcer and surrounding healthy skin.
  Other Names: Corneocyte evaluation

SUMMARY:
During a patient's hospital stay the skin can be exposed to forces from sitting or lying and attachment to different medical devices. Skin health is maintained healthy through regular movements to remove pressure from the skin surface. However, sometimes if the skin is exposed to loads for prolonged periods, it can be compromised, and red marks can appear (stage one pressure ulcer). In most cases, these changes in the skin can be recovered, through regular movement and nursing care. However, in a small number of cases, the skin damage can progress further until a wound appears. It is important to find out why this may occur, so that preventive strategies can be implemented to protect skin health. Therefore, the project focuses on evaluating changes in skin health following the development of a minor pressure ulcer (stage one).

This research proposal aims to better understand how the skin changes at the body sites compromised by stage 1 pressure ulcer, compared to healthy sites. This will be achieved via the use of measurements of skin health including physical sensors and sampling fluids and cells from the skin surface. The knowledge acquired from this study will help the understanding of how and why skin breaks down following early signs of damage. Some of the proposed sensing systems could then be used to support healthcare professionals to adopt the appropriate preventive strategies to avoid skin damage and subsequent wounds. A cohort of 50 patients will be recruited from a hospital setting, who present with a stage one pressure ulcer. Skin measurements will be taken three times to establish changes during their hospital stay. The investigators will establish if these measurements support the prediction of whether the stage one ulcer heals, remains the same, or progresses into a wound (stage two or higher pressure ulcer).

DETAILED DESCRIPTION:
This is a case controlled longitudinal observational study on patients who have the early signs of pressure ulcers, termed stage 1. In this study, a series of non-invasive measurements will be performed to assess skin status in individuals presenting with stage 1 pressure ulcers (PU). Photographic images of the compromised skin site of participants will also be collected. Participants will be tested using a well-established protocol, which consist of visiting the patient on three different occasions during their hospital stay. The first two visits will be on consecutive days while the third skin assessment session will be carried out a day before the patient is discharged. The investigator team will ensure that the sessions, which will last approximately 15-20 minutes, avoiding any interference with patients personal or healthcare commitments.

Different measurements on the participant skin surface will be taken using probes which are designed to monitor skin health (all probes are CE marked and have been employed previously in clinical trials). The measurements will include:

1. the pH (acidity) at the skin surface
2. the amount of water which is lost through the skin
3. skin hydration

In addition, sebum (oily substance) and cells from the compromised and healthy areas of the skin using commercial tapes were collected. The aforementioned skin parameters will be taken at each visit using non-invasive, harmless wireless probes, which will be placed gently in contact with the skin for a 1-minute duration. Each probe was cleaned in-between assessments following the NHS infection control policies. Skin sebum will also be taken at each assessment from the areas of interest using sebutapes, which will be gently applied to the skin for 2 minutes before removal. These commercially available tapes have been used extensively in dermatological research. Corneocytes (outermost surface cells) will be taken only on the first visit from both the compromised and healthy sites of the skin. This will be achieved using a harmless tape stripping technique during which standard sellotapes will be applied to the skin surface and slightly pressed for 5 seconds prior to removal.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years old
* Individuals of all genders and ethnicities
* Individuals presenting grade 1 PU (regardless of the anatomical location of the PU)
* Individuals admitted to UHST
* Have the capacity and English proficiency to provide informed consent

Exclusion Criteria:

* Individuals with broken skin
* Patients at end of life
* Patients who cannot be repositioned due to medical reasons
* Patients in COVID-19 areas
* Allergies or sensitivity to sebutape or Sellotape
* Current active skin condition on the areas of measurement
* Cognitive impairments which limit their ability to provide informed consent
* Inability to understand English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be purposefully sampled from a number of departments/units at University Hospital Southampton (UHS) Foundation Trust. According to information from the Tissue Viability Department, an average number of 50 patients are referred monthly with presentations of early signs of PUs. The study is designed to recruit 50 participants over a 12-month period
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Spatial and temporal differences in skin barrier function over a grade 1 pressure ulcer | 3 weeks.
  Case controlled differences in transepidermal water loss between the site of a grade 1 pressure ulcer and health adjacent skin. A Tewameter (CK, Germany) was used to assess skin barrier function sampled over a 30 second period. This was measured over the site of the grade 1 pressure ulcer and one that was 10cm lateral (healthy site). This outcome was measured in g/m2/hr.

SECONDARY OUTCOMES:
Spatial differences in skin corneocyte topography over a grade 1 pressure ulcer | 3 weeks.
  Case controlled differences in the maturity of corneocyte cells over a grade 1 pressure ulcer. Cells were collected from a PU-compromised site and an adjacent control area and their topographical properties were analysed. Atomic force microscopy (AFM) imaging and nanoindentation experiments were performed to assess topography.
Spatial differences in skin corneocyte maturity over a grade 1 pressure ulcer | 3 weeks.
  Case controlled differences in the maturity of corneocyte cells over a grade 1 pressure ulcer. Cells were collected from a PU-compromised site and an adjacent control area and maturation properties were analysed. Maturity of corneodesmosomes was indirectly measured by immunostaining of desmoglein-1 (Dsg1). Parameters of measurement included surface roughness Sq (nm) and Youngs Modulus of cells (MPa). Qualitative analysis of immunostaining of desmoglein-1 (Dsg1) was also included.
Spatial and temporal differences in skin inflammation over a grade 1 pressure ulcer | 3 weeks
  Case controlled differences in skin inflammatory biomarkers between the site of a grade 1 pressure ulcer and health adjacent skin. Sebutapes were collected over three sessions to investigate the temporal changes in the inflammatory response. The panel of cytokines investigated included high-abundance cytokines, namely, IL-1α and IL-1RA, and low abundance cytokines; IL-6, IL-8, TNF-α, INF-γ, IL-33, IL-1β and G-CSF. Spatial and temporal differences between sites were assessed and thresholds were used to determine the sensitivity and specificity of each biomarker. Concentrations of protein biomarkers in the sebum will be presented in picograms per ml.
Spatial and temporal differences in skin hydration over a grade 1 pressure ulcer | 3 weeks.
  Case controlled differences in skin hydration between the site of a grade 1 pressure ulcer and health adjacent skin. A Corneometer (CK, Germany) was used to assess skin hydration sampled 5 times over eac site. This was measured over the site of the grade 1 pressure ulcer and one that was 10cm lateral (healthy site). Stratum corneum hydration was measured in arbitrary units, according to the calibrated Corneometer.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Southampton (UHS) Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
As per University of Southampton and EU guidelines anonymised from the study can be accessed through our ePrints provider.

REFERENCES:
- [Background] Jayabal H, Abiakam NS, Filingeri D, Bader DL, Worsley PR. Inflammatory biomarkers in sebum for identifying skin damage in patients with a Stage I pressure ulcer in the pelvic region: A single centre observational, longitudinal cohort study with elderly patients. Int Wound J. 2023 Sep;20(7):2594-2607. doi: 10.1111/iwj.14131. Epub 2023 Mar 5. PMID 36872612
- [Result] Abiakam NS, Jayabal H, Filingeri D, Bader DL, Worsley PR. Spatial and temporal changes in biophysical skin parameters over a category I pressure ulcer. Int Wound J. 2023 Oct;20(8):3164-3176. doi: 10.1111/iwj.14194. Epub 2023 Apr 14. PMID 37060199
- See also: STINTS EU Marie Curie ITN funding home page — https://www.stints.eu/